CLINICAL TRIAL: NCT01890226
Title: A Mobile Personal Health Record for Behavioral Health Homes
Acronym: mPHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Druss, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00067447; 1R01MH100467-01 (NIH)
Record Dates: First submitted 2013-06-25; First posted 2013-07-01 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hypertension; Hyperlipidemia; Diabetes
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Experimental: Intervention (Experimental): Participants randomized to the intervention arm will receive the mobile personal health record.
  Interventions: Behavioral: Mobile Personal Health Record App.

INTERVENTIONS:
Behavioral: Mobile Personal Health Record App.
  Arms: Experimental: Intervention

SUMMARY:
Poor quality of medical care is a major contributor to excess medical morbidity and premature mortality in persons with serious mental illnesses (SMI). To address this problem, community mental health providers are increasingly partnering with safety net medical providers to develop behavioral health homes, integrated clinics in which persons with SMI receive coordinated medical and mental health care. However, behavioral health homes have faced logistical and privacy challenges in integrating electronic medical records across organizations.

This application proposes to develop and test a mobile Personal Health Record (mPHR) to overcome this problem while more fully engaging patients in their health care. The study will develop, test, and disseminate the mPHR. The investigators will develop the app building on experience and preliminary data from a PC-based PHR project, and link it to the medical and mental health EHR in a behavioral health home. Next, the investigators will conduct a randomized trial of the mPHR in 300 subjects randomized to the mPHR or usual care.

ELIGIBILITY:
Inclusion Criteria:

* one or more of the following conditions: hyperlipidemia, hypertension, diabetes
* able to give consent
* patient in the behavioral health home

Exclusion Criteria:

* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Druss, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Viewpoint Health & Oakhurst Medical Center, Conyers, Georgia, United States

REFERENCES:
- [Derived] Druss BG, Li J, Tapscott S, Lally CA. Randomized Trial of a Mobile Personal Health Record for Behavioral Health Homes. Psychiatr Serv. 2020 Aug 1;71(8):803-809. doi: 10.1176/appi.ps.201900381. Epub 2020 May 4. PMID 32362226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 311 participants were eligible and consented to participate.
Groups:
- Control: Control or usual care group: had access to the full array o services offered through the behavioral health homes.
- Experimental: Intervention: Participants randomized to the intervention arm will receive the mobile personal health record.
  Mobile Personal Health Record App.
Period: Overall Study
Arm/Group | Control | Experimental: Intervention
Started | 155 | 156
Completed | 155 | 156
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Control or usual care group: had access to the full array of services offered through the behavioral health homes.
- Total: Total of all reporting groups
Arm/Group | Control | Experimental: Intervention | Total
Number analyzed (Participants) | 155 | 156 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.54 (9.08) | 50.78 (8.45) | 50.66 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 95 | 187
  Male | 63 | 61 | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 29 | 58
  Black | 123 | 118 | 241
  Other Race | 3 | 9 | 12
Region of Enrollment [Number; unit: participants]
  United States | 155 | 156 | 311
total annual income [Count of Participants; unit: Participants]
  $0-$5,000 | 83 | 86 | 169
  $5,000-$10,000 | 43 | 42 | 85
  $10,000-$15,000 | 17 | 18 | 35
  More than $15,000 | 8 | 8 | 16
  Did not answer | 4 | 2 | 6
Medical Diagnosis [Count of Participants; unit: Participants]
  Diabetes | 68 | 68 | 136
  Heart Disease/CAD/CHD | 13 | 13 | 26
  Hyperlipidemia | 70 | 72 | 142
  Hypertension | 123 | 134 | 257
Mental Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 33 | 34 | 67
  Bipolar Disorder | 41 | 43 | 84
  Depression | 122 | 116 | 238
  Obsessive Compulsive Disorder | 6 | 4 | 10
  Post-Traumatic stress Disorder | 26 | 35 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Quality Score
Description: It is a measure of quality of care. The aggregate score represents the total number of eligible services received for an individual generated by dividing all instances in which recommended care was delivered by the number of times a participant was eligible for the indicator. The score ranges from 0 to 1 with higher scores indicating receipt of recommended care/services.
Time Frame: Baseline, 12 month post intervention
Population: Chart review data, which were used to assess overall quality of care, were available for all participants at baseline and 12-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental: Intervention
Number analyzed (Participants) | 155 | 156
score on a scale
  Baseline | 0.71 (0.12) | 0.70 (0.11)
  12-month post-baseline | 0.67 (0.16) | 0.70 (0.15)

2. Secondary Outcome: Change in Patient Assessment of Chronic Illness Care
Description: 20-item patient self-report instrument that assesses the extent to which patients with chronic illness report receiving care that aligns with the Chronic Care Model. The summary score ranges from 1 to 5 with a higher score indicating patient's perception of greater involvement in self-management and receipt of chronic care counseling.
Time Frame: Baseline, 6 month post intervention, 12 month post intervention
Population: Completion rates for patient interviews were 91.9% at 6-months and 84.6% for 12 months, with similar rates of attrition in both groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental: Intervention
Number analyzed (Participants) | 155 | 156
score on a scale
  Baseline | 3.23 (1.00) | 3.20 (0.95)
  6-month post-baseline: number analyzed (Participants) | 141 | 145
  6-month post-baseline | 3.32 (1.01) | 3.32 (0.93)
  12-month post-baseline: number analyzed (Participants) | 131 | 132
  12-month post-baseline | 3.18 (0.95) | 3.25 (0.94)

3. Secondary Outcome: Change in Patient Activation Measure
Description: Assesses a patients' perceived ability to manage their illnesses and their healthcare visits. Patient Activation Measure Scores were summed to calculate the overall raw score then transformed to an activation scale ranging from 0 to 100. Higher scores indicate greater patient activation.
Time Frame: Baseline, 6 month post intervention, 12 month post intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental: Intervention
Number analyzed (Participants) | 155 | 156
score on a scale
  Baseline | 57.83 (13.65) | 58.78 (14.65)
  6-month post-baseline: number analyzed (Participants) | 141 | 145
  6-month post-baseline | 60.88 (15.18) | 59.82 (15.89)
  12-month post-baseline: number analyzed (Participants) | 132 | 132
  12-month post-baseline | 32.08 (14.77) | 61.61 (16.19)

4. Secondary Outcome: Change in Health-related Quality of Life
Description: Measured using the Physical and Mental Component Summary scales of the SF-12. Assesses a patients' perceived health related quality of life.
  The composite physical (PCS) and mental component (MCS) summary scores for the SF-12 are each scored on a 0-100 scale. Higher scores indicate better functioning.
Time Frame: Baseline, 6 month post intervention, 12 month post intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental: Intervention
Number analyzed (Participants) | 150 | 147
score on a scale
  SF-12 PCS Baseline | 35.70 (11.62) | 35.74 (11.83)
  SF-12 PCS 6-month: number analyzed (Participants) | 133 | 138
  SF-12 PCS 6-month | 36.32 (11.52) | 37.20 (11.94)
  SF-12 PCS 12-month: number analyzed (Participants) | 130 | 129
  SF-12 PCS 12-month | 36.09 (11.75) | 37.03 (12.15)
  SF-12 MCS Baseline | 36.55 (13.25) | 35.50 (12.54)
  SF-12 MCS 6-month: number analyzed (Participants) | 133 | 138
  SF-12 MCS 6-month | 38.70 (13.18) | 39.16 (13.48)
  SF-12 MCS 12-month: number analyzed (Participants) | 130 | 129
  SF-12 MCS 12-month | 41.16 (11.61) | 41.68 (14.04)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Serious and non serious adverse events that were reported during the 12 months follow up time.
Arm/Group | Control | Experimental: Intervention
All-Cause Mortality (participants affected / at risk) | 1/155 | 3/156
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/156
Other Adverse Events (participants affected / at risk) | 0/155 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT01890226/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT01890226/ICF_001.pdf